CLINICAL TRIAL: NCT03332329
Title: Efficacy and Safety of Combination Therapy With Entecavir, Peginterferon Alfa-2b and Immunomodulators in Nucleoside or Nucleotide Analogue (NA)-Suppressed Chronic Hepatitis B Patients
Brief Title: Sequential/Combination Therapy in Nucleoside or Nucleotide Analogue (NA)-Suppressed Chronic Hepatitis B Patients
Acronym: NPGV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Prof, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPGV study
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis b
Keywords: HBsAg; PegIFN; ETV; Chronic Hepatitis B (CHB); HBV; GMCSF
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Granulocyte-Macrophage Colony-Stimulating Factor; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential combination arm (Experimental): Drug: Entecavir for 60 weeks Drug: HBV vaccine (60ug/month, every four weeks) for 24 weeks Drug: Granulocyte Macrophage Colony Stimulating Factor (75 μg/day, first 5 days each month, subcutaneous) from baseline to week 16 and from week 60 to week 84 Drug: Y peginterferon alfa-2b (180 μg/week, subcutaneous) from week 16 to week 108
  Interventions: Drug: Entecavir; Drug: Granulocyte Macrophage Colony Stimulating Factor; Drug: Y peginterferon alfa-2b; Drug: HBV vaccine

INTERVENTIONS:
Drug: Entecavir — Entecavir is used for 96 weeks
  Other Names: ETV
Drug: Granulocyte Macrophage Colony Stimulating Factor — Granulocyte-macrophage colony stimulating factor is used intermittently from baseline to week 16 and from 60 to week 84
  Other Names: GMCSF
Drug: Y peginterferon alfa-2b — Y peginterferon alfa-2b is used for 96 weeks
  Other Names: peginterferon a-2b
Drug: HBV vaccine — 60ug HBV vaccine is used every four week for 24 weeks
  Other Names: vaccine

SUMMARY:
The aim of the prospective study is to determine whether combination/ sequential therapy with Entecavir, Peginterferon alfa-2b and immunomodulators Granulocyte Macrophage Colony Stimulating Factor (GMCSF)+vaccine could induce HBsAg loss in chronic hepatitis B patients with maintained Hepatitis B Virus (HBV) DNA suppression on long-term nucleoside or nucleotide analogue (NA).

DETAILED DESCRIPTION:
Patents who were treated with NA at least one year and achieved HBV DNA suppression are enrolled in this study, they will receive Entecavir (ETV) for 60 weeks, HBV vaccine (60ug/month, every four weeks) for 24 weeks, GMCSF (75 μg/day, first 5 days each month, subcutaneous) from baseline to week 16 and from week 60 to week 84, and Y peginterferon alfa-2b (180 μg/week, subcutaneous) from week 16 to week 108.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. HBsAg positive, entecavir and or adefovir dipivoxil are used at least 1 year including patients with nucleotides or nucleoside resistance history;
3. Before nucleotides or nucleosides treatment, ALT > 2 upper limit of normal value (ULN), HBV DNA >10000 copies/ml, HBsAg positive;
4. Serum HBV DNA < 1000 copies/ml;
5. 2000 IU/ml ≤HBsAg≤6000 IU/ml;
6. HBsAg positive;
7. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug;
8. Absence of cirrhosis confirmed by ultrasonic test;
9. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. Patients who had NAs resistance and HBV DNA > 1000 copies/ml, or treatment of drugs with interferon longer than 6 months;
2. Other antiviral, anti-neoplastic or immunomodulatory treatment (including supra physiologic doses of steroids and radiation) 6 months prior to the first dose of randomized treatment (except for 7 days of acyclovir for herpetic lesions more than 1 month prior to first administration of randomized treatment). Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation are also excluded;
3. Women with ongoing pregnancy or breast-feeding;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D(Those hospitals which have the ability to do the test will do) and/or human immunodeficiency virus (HIV);
5. ALT >10 ULN;
6. Evidence of decompensated liver disease (Child-Pugh score > 5). Child-Pugh > 5 means, if one of the following 5 conditions are met, the patient has to be excluded:
7. one of the following 5 conditions are met, the patient has to be excluded:
8. Serum albumin < 3.5 g/L;
9. Prothrombin time > 3 seconds prolonged;
10. Serum bilirubin > 34 µ mol/L;
11. History of encephalopathy;
12. History of variceal bleeding;
13. Ascites;
14. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
15. Signs or symptoms of hepatocellular carcinoma, patients with a value of alpha-fetoprotein > 100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months. Patients with values < 20 ng/mL but > 100 ng/mL may be enrolled, if hepatic neoplasia has been excluded by liver imaging;
16. Neutrophil count < 1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening;
17. Hemoglobin < 11.5 g/dL for females and <12.5 g/dL for men;
18. Serum creatinine level > 1.5 ULN in screening period.
19. Phosphorus < 0.65 mmol/L;
20. antinuclear antibody (ANA) > 1:100;
21. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
22. History of a severe seizure disorder or current anticonvulsant use;
23. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
24. History of chronic pulmonary disease associated with functional limitation;
25. Diseases that interferon and Nucleotides or nucleosides are not suitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAg loss rate | at week 108
  Percentages of patients who achieve HBsAg loss at the end of treatment

SECONDARY OUTCOMES:
HBsAg level | at week 60
  Dynamic change in HBsAg level from baseline to the end of treatment
HBsAg level | at week 108
  Dynamic change in HBsAg level from baseline to the end of treatment
decline in HBsAg level | at week 60
  Decline in HBsAg level from baseline to the end of treatment
decline in HBsAg level | at week 108
  Decline in HBsAg level from baseline to the end of treatment
HBsAb appearance rate | at week 108
  Percentages of HBsAb appearance at the end of treatment
HBsAb seroconversion rate | at week 108
  Percentages of HBsAb seroconversion at the end of treatment
HBeAg loss rate | at week 108
  Percentages of HBeAg loss in the HBeAg-positive patients at the end of treatment
HBeAg seroconversion rate | at week 108
  Percentages of HBeAg seroconversion in the HBeAb-negative patients at the end of treatment
Rate of HBV DNA level <1000 copies/mL | at week 108
  Percentages of HBV DNA level <1000 copies/mL at the end of treatment
Rate of alanine aminotransferase (ALT) normalisation | at week 108
  Percentages of ALT normalisation at the end of treatment
Sustained HBsAg loss rate | at week 156
  Percentages of sustained HBsAg loss at the end of follow-up
The rate of progression to cirrhosis | at week 156
  The rate of progression to cirrhosis at the end of follow-up
The incidence rate of hepatocarcinoma | at week 156
  The incidence rate of hepatocarcinoma at the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Undecided